CLINICAL TRIAL: NCT06328062
Title: Comparison Efficacy of Mirogabalin and Pregabalin in Total Knee Arthroplasty. a Randomized Controlled Trial
Brief Title: Comparing Efficiency of Mirogabalin and Pregabalin in Primary TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Principle investigator, Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUH Mirogabalin TKA
Record Dates: First submitted 2024-03-08; First posted 2024-03-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Pain Postoperative; Osteoarthritis; Total Knee Arthroplasty
Keywords: mirogabalin; pregabalin; pain postoperative; TKA
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis | interventions — mirogabalin; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirogabalin (Experimental): Participants will receive 5 mg of mirogabalin, taken as half a tablet, every day twice a day, after breakfast and dinner, for 6 weeks.
  Interventions: Drug: Mirogabalin
- Pregabalin (Active Comparator): Participants will receive 50 mg of pregabalin, taken as a tablet, every day twice a day, after breakfast and dinner, for 6 weeks.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Mirogabalin — Participants will receive 5 mg of mirogabalin, taken as half a tablet, every day twice a day, after breakfast and dinner, for 6 weeks.
  Arms: Mirogabalin
Drug: Pregabalin — Participants will receive 50 mg of pregabalin, taken as a tablet, every day twice a day, after breakfast and dinner, for 6 weeks.
  Arms: Pregabalin

SUMMARY:
The goal of this RCT is to compare efficacy between mirogabalin and pregabalin in pain reducing after unilateral primary total knee arthroplasty.

The main question[s] it aims to answer are:

• Does mirogabalin have better pain reduction than pregabalin after unilateral primary total knee arthroplasty.

Participants will randomized to mirogabalin or pregabalin group and will take the drug for 6 weeks after TKA. Researchers will compare to pregabalin group to see pain and functional outcomes after TKA.

DETAILED DESCRIPTION:
After surgery is complete, you will be randomly assigned to receive painkillers Mirogabalin or Pregabalin along with other standard medications.

Surgery by Mirogabalin group: Participants received 5 mg of mirogabalin, taken as half a tablet, every day.

Twice a day, after breakfast and dinner, for 6 weeks. In the pregabalin group: Participants received 50 mg of pregabalin, one tablet taken daily.

Twice a day, after breakfast and dinner, for 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-85 years old
2. Unilateral primary osteoarthritis undergoing primary TKA
3. ASA I-III

Exclusion Criteria:

1. GFR <60
2. Allergy to drug in this study
3. Cannot underwent spinal anesthesia and adductor canal block
4. Taking gabapentinoid within 3 months before surgery
5. History of previous knee surgery
6. Severe liver disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | Every 6 hours after surgery for 2 days, then twice a day for 2 weeks, then once a week until 12 week after surgery.
  Visual analog scale at rest and motion (0-100 points, 0 mean best, 100 mean worst)

SECONDARY OUTCOMES:
Morphine consumption | 72 hours after surgery
  Total morphine consumption in hospital (mg)
Range of motion | 24 hour, 48 hour, 2 week, 6 week and 12 week after surgery
  Using long arm goniometer (degrees)
Knee society score | 2 week, 6 week and 12 week after surgery
  report in point (0-100, 0 mean worst, 100 mean best)
Knee injury and Osteoarthritis Outcome Score (KOOS) | 2 week, 6 week and 12 week after surgery
  report in point (0-100, 0 mean worst, 100 mean best)
Sedation score | 24 hour, 48 hour, 2 week, 6 week and 12 week after surgery
  report in point (0-100, 0 mean best, 100 mean worst)
Incidence of Somnolence and dizziness | everyday until 14 days then once a week until 12 weeks after surgery
  Using scale "Mild, moderate and severe"
Total hospital stay | up to 1 week
  Number of days the patient stays for surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hannon CP, Fillingham YA, Browne JA, Schemitsch EH, Mullen K, Casambre F, Visvabharathy V, Hamilton WG, Della Valle CJ. The Efficacy and Safety of Gabapentinoids in Total Joint Arthroplasty: Systematic Review and Direct Meta-Analysis. J Arthroplasty. 2020 Oct;35(10):2730-2738.e6. doi: 10.1016/j.arth.2020.05.033. Epub 2020 May 26. PMID 32586656
- [Background] Kim JY, Abdi S, Huh B, Kim KH. Mirogabalin: could it be the next generation gabapentin or pregabalin? Korean J Pain. 2021 Jan 1;34(1):4-18. doi: 10.3344/kjp.2021.34.1.4. PMID 33380563